CLINICAL TRIAL: NCT02516345
Title: Randomized Controlled Trial of an Incentive-based Physical Activity Program Targeting Both Children and Adults (FIT-FAM)
Acronym: FIT-FAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSRG13may010
Record Dates: First submitted 2015-04-27; First posted 2015-08-05 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Physical Activity
Keywords: Physical activity; Financial incentives; Children; Parents; RCT; Wireless pedometer
MeSH Terms: conditions — Motor Activity | interventions — Fertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Child-based Incentive (CBI) (Active Comparator): Children earn rewards each week (with the week beginning on Monday and ending on Sunday) that they log 10,000 daily steps on the Fitbit according to the schedule below and their matched parent logs at least 2,000 steps on ≥4 of 7 days each week (regardless of which 4 of the 7 days they wear it). Incentives are tied, in addition to child's activity, to parent's Fitbit wear so that the investigators are better able to capture parent's activity in this arm.
  Step Targets for Children in CBI arm:
  * Months 1 - 3: ≥10,000 daily steps on ≥4 out of 7 days each week
  * Months 4 - 6: ≥10,000 daily steps on ≥5 out of 7 days each week
  * Months 7 - 12: ≥10,000 daily steps on ≥6 out of 7 days each week
  Interventions: Device: Fitbit; Behavioral: Incentives
- Family-based Incentive (FBI) (Experimental): Children earn rewards each week that they log daily steps on the Fitbit according to the schedule below but only if their matched parent also logs 10,000 steps according to the schedule below. Otherwise, children earn no incentive for that week.
  Step targets for children and parents in FBI arm:
  * Months 1 - 3: ≥10,000 daily steps on ≥4 out of 7 days each week
  * Months 4 - 6: ≥10,000 daily steps on ≥5 out of 7 days each week
  * Months 7 - 12: ≥10,000 daily steps on ≥6 out of 7 days each week
  Interventions: Device: Fitbit; Behavioral: Incentives

INTERVENTIONS:
Device: Fitbit — Fitbit devices are wireless pedometers that track the steps of participants, and will be offered in conjunction with a tailored website with customized information for participants.
  Other Names: Fitbit Zip, Fitbit Flex, wireless pedometer, physical activity tracker
Behavioral: Incentives — Incentives will be awarded to participating children for meeting step targets as measured by the Fitbit pedometer.
  Other Names: Rewards, gift vouchers

SUMMARY:
This study aims to test whether incentives can motivate children to promote increased physical activity of a working parent while also increasing their own activity levels.

DETAILED DESCRIPTION:
There is overwhelming evidence that sustained physical activity reduces the risk of many common diseases. Yet, data reveal low levels of physical activity among working age adults and their children in Singapore. One strategy that has been successfully employed to influence behaviours of parents is to use their children as an intermediary. This strategy has a successful track record in public health, where children have helped their parents quit smoking and wear seatbelts.

In this study, the investigators propose to test whether children can promote increased physical activity of a working parent at the same time that they increase their own activity level. This proposal is an extension of a prior study where the investigators showed that modest financial incentives can increase physical activity levels among children. The investigators now propose to conduct a follow-on trial where the reward is tied not only to the child's own steps, but to that of a parent. Rewards will be based on step activity measured through a state-of-the-art wireless step counter worn on the wrist or hip. Just as children were motivated to increase their own activity levels in efforts to achieve the incentive, the investigators hypothesize that they will also be effective advocates for increasing the activity levels of their parents.

Specifically, the investigators propose to conduct a 12 month two-arm randomized controlled trial (RCT) to evaluate the efficacy of the family based incentive scheme on working parents' physical activity as measured via accelerometry. The investigators hypothesize that parents in the family-based incentive arm (FBI) will show a greater number of daily steps at the interim 6 month assessment and the final 12 month assessment point compared to parents in the child based incentive (CBI) arm, as measured by accelerometry. Secondary aims test the effects of the intervention on parent's and child's MVPA bout minutes per week, MVPA minutes, and other physical activity endpoints measured by accelerometry, child's steps, parent's and child's activity levels throughout the intervention period measured by the pedometer, and on health outcomes and health-related quality of life of parents at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Child must be aged 7 - 11 years
* Parent must be aged 25 - 65 years
* Parent must be full-time employee at the time of enrolment
* Parent should be Singaporean citizen or permanent resident
* Parent and child must provide at least 4 valid days of accelerometer data (3 weekday days and 1 weekend day of at least 10 hours of wear time each day)

Exclusion Criteria:

* Difficulty walking up 10 stairs without stopping (for parents)
* Having any medical condition that may limit their ability to walk as a means of physical activity (for parents)
* Pregnant (for parents)
* Are unwilling to wear a wireless pedometer for 12 months (for parents and children)
* Are unwilling to wear an accelerometer for 1 week at baseline, month 6, and month 12 assessments (for parents and children)

Conditional Eligibility Criteria:

If parents meet the following criteria, they will be required to provide an approval note from a physician to be able to participate in the study-

* Self-reported medical conditions such as hypertension or diabetes that limit the ability to walk
* Answer 'YES' to any Physical Activity Readiness (PAR-Q) question
* Family history of heart conditions
* BMI>40kg/m2
* Children on whose behalf parents answer 'YES' to any PAR-Q question will be permitted to enrol only if they provide written approval from a medical doctor

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-06-03 (Actual)

PRIMARY OUTCOMES:
Changes in step count of parents from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Step counts of parents will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.

SECONDARY OUTCOMES:
Changes in step count of children from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Step counts of children will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in moderate to vigorous physical activity (MVPA) bout minutes of parents from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  MVPA will be assessed via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, 6 months, and 12 months. MVPA bout minutes are defined as a total of 10 or more consecutive minutes above the vector magnitude cutoff point of 2690 counts per min, with allowance for interruptions of 1-2 min at a magnitude less than the cutoff point.
Changes in moderate to vigorous physical activity (MVPA) bout minutes of children from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  MVPA will be assessed via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, 6 months, and 12 months. MVPA bout minutes are defined as a total of 10 or more consecutive minutes above the vector magnitude cutoff point of 2690 counts per min, with allowance for interruptions of 1-2 min at a magnitude less than the cutoff point.
Changes in moderate to vigorous physical activity (MVPA) minutes of parents from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Total MVPA minutes (including those not in bouts of 10 minutes) during each assessment period at baseline, month 6, and month 12. This will be assessed via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day).
Changes in moderate to vigorous physical activity (MVPA) minutes of children from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Total MVPA minutes (including those not in bouts of 10 minutes) during each assessment period at baseline, month 6, and month 12. This will be assessed via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day).
Changes in total volume of physical activity of parents from baseline to month 6 and month 12. | Baseline, 6 months and 12 months
  Average daily volume of physical activity will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in total volume of physical activity of children from baseline to month 6 and month 12. | Baseline, 6 months and 12 months
  Average daily volume of physical activity will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in sedentary behaviour of parents from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Average daily minutes of sedentary behaviour will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in sedentary behaviour of children from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Average daily minutes of sedentary behaviour will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in light minutes of parents from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Average daily light minutes will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in light minutes of children from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Average daily light minutes will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in total moderate minutes of parents from baseline to month 6 and month 12. | Baseline, 6 months and 12 months
  Average daily moderate minutes will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in total moderate minutes of children from baseline to month 6 and month 12. | Baseline, 6 months and 12 months
  Average daily moderate minutes will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in total vigorous minutes of parents from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Average daily vigorous minutes will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in total vigorous minutes of children from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Average daily vigorous minutes will be measured via the ActiGraph GT-3X+ accelerometer worn for a one-week period (with a minimum of 3 weekday days and 1 weekend day of at least 10 hours of wear time each day) at baseline, month 6, and month 12.
Changes in daily average steps of parents over the 12 month study duration. | Daily from months 1 - 12
  Daily average steps will be calculated based on data captured by the Fitbit wireless pedometer.
Changes in daily average steps of children over the 12 month study duration. | Daily from months 1 - 12
  Daily average steps will be calculated based on data captured by the Fitbit wireless pedometer.
Changes in percentage of parents meeting weekly step targets over the 12 month study duration. | Daily from months 1 - 12
  Percentage meeting weekly step targets will be calculated based on data captured by the Fitbit wireless pedometer.
Changes in percentage of children meeting weekly step targets over the 12 month study duration. | Daily from months 1 - 12
  Percentage meeting weekly step targets will be calculated based on data captured by the Fitbit wireless pedometer.
Changes in percentage of parent-child dyads meeting weekly step targets over the 12 month study duration. | Daily from months 1 - 12
  Percentage meeting weekly step targets will be calculated based on data captured by the Fitbit wireless pedometer.
Change in weight of parents from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  Weight of parents will be measured at baseline, month 6, and month 12, and the difference will be calculated.
Change in systolic blood pressure of parents from baseline to month 6 and month 12. | Baseline, 6 months and 12 months
  Systolic blood pressure of parents will be measured at baseline, month 6, and month 12, and the difference will be calculated.
Change in cardiorespiratory fitness of parents from baseline to month 6, and month 12. | Baseline, 6 months and 12 months
  VO2max of parents will be measured at baseline, month 6, and month 12, and the difference will be calculated.
Change in health-related quality of life of parents from baseline to month 6, and month 12. | Baseline, months and 12 months
  Health-related quality of life of parents at baseline, month 6, and month 12 will be measured via the EQ-5D-5L questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore

REFERENCES:
- [Derived] Finkelstein EA, Lim RSM, Ward DS, Evenson KR. Leveraging family dynamics to increase the effectiveness of incentives for physical activity: the FIT-FAM randomized controlled trial. Int J Behav Nutr Phys Act. 2020 Sep 10;17(1):113. doi: 10.1186/s12966-020-01018-2. PMID 32912260